CLINICAL TRIAL: NCT01382030
Title: A Phase II Study Evaluating Neo-/Adjuvant EIA Chemotherapy, Surgical Resection and Radiotherapy in High-risk Soft Tissue Sarcoma
Brief Title: Neoadjuvant and Adjuvant Chemotherapy in High-risk Soft Tissue Sarcoma
Acronym: NeoWTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: PD Dr. med. Gerlinde Egerer, Department of Hematology, Heidelberg University Clinics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-002501-72; 2004-002501-72 (EudraCT Number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; High-risk; Neoadjuvant; Adjuvant; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): All patients receive 4 cycles of EIA chemotherapy pre- and postoperatively. There is no further observation arm. The study is non-randomized.
  Interventions: Drug: EIA chemotherapy

INTERVENTIONS:
Drug: EIA chemotherapy — ifosfamide 1500 mg/m² iv days 1 - 4, etoposide 125 mg/m² iv days 1 and 4, and adriamycin 50 mg/m² iv day 1

SUMMARY:
Neo- and adjuvant chemotherapy is used in high-risk soft tissue sarcoma to improve systemic control. Patients in this trial are treated with 4 cycles of chemotherapy (EIA, etoposide, ifosfamide, adriamycin) preoperatively, followed by local surgery and radiotherapy. An additional 4 cycles of adjuvant chemotherapy is administered. Treatment response is assessed by MRI and CT scans and FDG-PET in a subgroup of patients.

DETAILED DESCRIPTION:
The role of chemotherapy in high-risk soft tissue sarcoma is controversial. Though many patients undergo initial curative resection, distant metastasis is a frequent event resulting in 5-year overall survival rates of only 50 - 60%. Neo-adjuvant and adjuvant chemotherapy has been applied to achieve pre-operative cytoreduction, assess chemosensitivity and to eliminate occult metastasis. The current protocol comprises for cycles of neoadjuvant chemotherapy ((EIA, etoposide 125 mg/m2 iv days 1 and 4, ifosfamide 1500 mg/m2 iv days 1 - 4, doxorubicin 50 mg/m2 day 1, pegfilgrastim 6 mg sc day 5), local surgery and radiotherapy as well as further 4 cycles of adjuvant EIA. Treatment response is assessed by MRI and CT scans and FDG-PET in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Soft tissue sarcoma histology
* Tumor size >= 5 cm
* Deep/extracompartimental localization
* Grade 2/3 (FNCLCC)
* Patients with inadequate previous therapy
* Age 18-65 years
* normal bone marrow function
* normal liver function
* normal renal function
* Karnofsky index >=80%

Exclusion Criteria:

* Chordoma
* Chondrosarcoma
* Kaposi´ sarcoma
* Neuroblastoma
* Mesothelioma
* Osteosarcoma/Ewings´sarcoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years after study completion
  Disease-free survival will be calculated from the time of definite surgery to radiologically proven local or distant failure or patient´s death due to sarcoma related cause.

SECONDARY OUTCOMES:
Overall Survival | 2 years after study completion
  Overall survival will be calculated as the time interval from the date of therapy induction to patient's death or last follow up.
Grade of histological necrosis | After definite surgery, approx. 12-15 weeks after study inclusion
  Grade of histological necrosis in tumor specimen will be assessed after surgery and graded according to Salzer-Kuntschik.
Hematological toxicity | Once weekly for an average of 8 months
  Hematological toxicity will be assessed by complete blood counts. Toxicity will be graded according to CTCAE.
Renal Toxicity | Once weekly for an average of 8 months
  Renal toxicity will be assessed by changes from baseline creatinin levels. Toxicity will be graded according to CTCAE.
Liver Toxicity | Once weekly for an average of 8 months
  Liver toxicity will be assessed by changes from baseline liver function tests, e.g. ASAT/ALAT. Toxicity will be graded according to CTCAE.
Correlation of Tumor Necrosis and Decline in PET SUV | After tumor resection, approx. 12-15 weeks after study inclusion
  Decline in PET SUV will be correlated with grade of histological necrosis in tumor specimen after surgery.
Cardiac Toxicity | Every 6 weeks for an average of 8 months
  Changes in cardiac ejection fraction will be assessed by echocardiograms. Toxicities will be graded according to CTCAE.
Radiologic Tumor Response | Every 6 weeks for an average of 8 months, then every 3 months for 2 years
  Tumor response to therapy will be assessed by MRI and CT scans. Response will graded according to RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gerlinde Egerer, MD, Principal Investigator — Department of Hematology, Heidelberg University Clinics
Locations (1):
- Heidelberg University Clinics, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Roeder F, Lehner B, Schmitt T, Kasper B, Egerer G, Sedlaczek O, Grullich C, Mechtersheimer G, Wuchter P, Hensley FW, Huber PE, Debus J, Bischof M. Excellent local control with IOERT and postoperative EBRT in high grade extremity sarcoma: results from a subgroup analysis of a prospective trial. BMC Cancer. 2014 May 20;14:350. doi: 10.1186/1471-2407-14-350. PMID 24885755
- [Derived] Schmitt T, Lehner B, Kasper B, Bischof M, Roeder F, Dietrich S, Dimitrakopoulou-Strauss A, Strauss LG, Mechtersheimer G, Wuchter P, Ho AD, Egerer G. A phase II study evaluating neo-/adjuvant EIA chemotherapy, surgical resection and radiotherapy in high-risk soft tissue sarcoma. BMC Cancer. 2011 Dec 7;11:510. doi: 10.1186/1471-2407-11-510. PMID 22152120